CLINICAL TRIAL: NCT02128698
Title: Physical Activity and Protein Supplementation After Bariatric Surgery
Brief Title: Physical Activity and Protein Supplementation After Bariatric Surgery (PAPAB)
Acronym: PAPAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hohenheim (Other)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ZEM_Minigrad_CH
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Bariatric Surgery Candidate
Keywords: Bariatric surgery; Protein supplementation; Physical activity; Muscle mass; Weight loss; Physical fitness; Muscle strength
MeSH Terms: conditions — Motor Activity; Weight Loss | interventions — Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Protein and computer-assisted exercise (Experimental): Patient group which takes daily protein supplements and is advised to do exercise 4 times per week by using Nintendo Wii Balance Board and Wii Fit Plus Software during 6 months after bariatric surgery.
  Interventions: Dietary Supplement: Protein; Behavioral: Computer-assisted exercise
- Placebo and computer-assisted exercise (Placebo Comparator): Patient group which takes daily control product and is advised to do exercise 4 times per week by using Nintendo Wii Balance Board and Wii Fit Plus Software during 6 months after bariatric surgery.
  Interventions: Dietary Supplement: Placebo; Behavioral: Computer-assisted exercise
- Protein and usual exercise (Active Comparator): Patient group which takes daily protein supplements and is advised to do exercise 4 times per week by using written exercise instructions during 6 months after bariatric surgery.
  Interventions: Dietary Supplement: Protein; Behavioral: Usual exercise
- Placebo and usual exercise (Active Comparator): Patient group which takes daily control product and is advised to do exercise 4 times per week by using written exercise instructions during 6 months after bariatric surgery.
  Interventions: Dietary Supplement: Placebo; Behavioral: Usual exercise

INTERVENTIONS:
Dietary Supplement: Protein — Postoperative intake of 25 g per day starting on the first day after hospital discharge until 6 months postoperatively.
  Other Names: Resource Instant Protein 88, Néstle Health Nutrition
  Arms: Protein and computer-assisted exercise; Protein and usual exercise
Dietary Supplement: Placebo — Postoperative intake of 25 g per day starting on the first day after hospital discharge until 6 months postoperatively.
  Other Names: Resource Maltodextrin, Néstle Health Nutrition
  Arms: Placebo and computer-assisted exercise; Placebo and usual exercise
Behavioral: Computer-assisted exercise — Postoperative regular computer-assisted exercise using Nintendo Wii Mini, Nintendo Wii Balance Board and Wii Fit Plus Software. Exercise is advised to be done 4 times per week.
  Arms: Placebo and computer-assisted exercise; Protein and computer-assisted exercise
Behavioral: Usual exercise — Postoperative regular exercise using written exercise instructions. Exercise is advised to be done 4 times per week.
  Arms: Placebo and usual exercise; Protein and usual exercise

SUMMARY:
The purpose of this study is to determine wether regular physical activity in combination with protein supplementation after bariatric surgery can reduce the loss of muscle mass and wether a computer-assisted exercise program is more effective than a usual exercise program regarding frequency of physical activity, fitness and muscular strength.

DETAILED DESCRIPTION:
Bariatric surgery has become a major treatment option for severe obesity in adults. Despite the advantages of bariatric surgery, attention needs to be paid to the possible risks following the surgical treatment. Postoperative risks include protein deficiency and pronounced muscle mass loss. Indeed, numerous studies indicate a significant reduction in lean body mass resulting from protein deficiency after bariatric surgery.

Dietary proteins have shown to play an important role in body weight regulation. A protein-rich diet attains satiety and thereby facilitates reduction in overall energy intake. It has also shown to enhance food-induced thermogenesis. Furthermore, a protein-rich diet - ideally in combination with exercise - preserves lean body mass and thus resting energy expenditure leading to an improvement of long-term energy balance. Therefore, protein-rich diets or protein supplements, respectively, might facilitate weight loss, especially body fat loss and protect against loss in muscle mass in patients who underwent bariatric surgery. The aim of the present randomized, placebo-controlled, double blind pilot study was to test the possible benefit of proteins in combination with exercise in patients undergoing bariatric surgery, and to examine, whether computer-assisted exercise is advantageous when comparing it to a usual exercise program using written exercise instructions. Therefore, we study the influence of postoperative protein supplementation in combination with computer-assisted exercise on body composition changes, and body weight reduction, as well as physical fitness, protein status and muscle function in obese patients after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 - 65 years
* Body weight of ≤ 150 kg
* BMI > 35 kg/m2
* Indication for laparoscopic sleeve gastrectomy and laparoscopic Roux-en-Y gastric bypass. The decision about the type of surgery is performed independent of the study by the surgeons in charge according to the German S3 guideline.

Exclusion Criteria:

* Kidney diseases of any kind
* Serious gastrointestinal diseases (e.g. Morbus Crohn, Colitis Ulcerosa, etc.)
* Serious musculoskeletal diseases
* Serious heart diseases (Myocardial infarction, stent implantation, stroke, etc.)
* Intake of blood thinning medicine (e.g. ASS, Marcumar, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Lean body mass loss expressed as percentage of weight loss [%] | At month 6
  Lean body mass is measured by using body impedance analysis. The content of lean body mass in lost weight is calculated using the lost weight in kg and the lost lean body mass in kg.

SECONDARY OUTCOMES:
Relative weight loss [%] | At month 6
Grip strength [lb] | At month 6
  Grip strength [lb] is measured by using a hydraulic force measuring device.
Grip strength endurance [sec] | At month 6
  Grip strength endurance [sec] is measured by using a hydraulic force measuring device.
Physical fitness [repetitions per 30 sec] / [distance in meters] | At month 6
  Physical fitness is assessed by the "30 Second Sit to Stand Test" and the "6 Minute Walk Test (6MWT)". The results of these tests are stated as repetitions per 30 seconds, and distance in meters, respectively.

OTHER OUTCOMES:
Blood proteins | At month 6
  Blood proteins, including albumin, prealbumin, transferrin, and total protein, are measured to assess blood protein status.
Urea and creatinine excretion | At month 6
  Urea and creatinine excretion are measured in 24 h urine samples.
Frequency of exercise | During the whole study period of 6 months
  The frequency of exercise is assessed by using heart rate monitors, which are able to save all exercise data of the patients.
Health related quality of life | At month 6
  Health related quality of life is assessed by using the standardized questionnaire "short form 36" (SF36).
Body weight related quality of life | At month 6
  Body weight related quality of life is assessed by using the standardized questionnaire "Impact of Weight on Quality of Life" (IWQOL).
Outcome after bariatric surgery | At month 6
  Outcome is measured by using the standardized instrument "Bariatric Analysis and Reporting Outcome System" (BAROS) which considers excess weight loss, improvement of obesity-related comorbidities, and health related quality of life.
Anxiety disorder | At month 6
  Anxiety is assessed by using the standardized questionnaire "Generalised Anxiety Disorder Assessment" (GAD7).
Mental health | At month 6
  Mental health is assessed by using the standardized questionnaire "Patient Health Questionnaire" (PHQ9).

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Königsrainer, Professor, Study Director — Department of General, Visceral, and Transplant Surgery, University Hospital of Tübingen, Tübingen, Germany; Tobias Meile, MD, Principal Investigator — Department of General, Visceral, and Transplant Surgery, University Hospital of Tübingen, Tübingen, Germany; Stephan C Bischoff, Professor, Study Chair — Department of Nutritional Medicine, University of Hohenheim, Stuttgart, Germany
Locations (1):
- Department of General, Visceral, and Transplant Surgery, University Hospital of Tübingen, Tübingen, Germany